CLINICAL TRIAL: NCT06424444
Title: A Multicenter, Phase 3, Randomized, Double-Masked, Parallel-Group, Vehicle-Controlled, Environment Exposure Clinical Trial to Assess the Efficacy and Safety of 0.25% Reproxalap Ophthalmic Solution Compared to Vehicle in Subjects With Dry Eye Disease
Brief Title: A Clinical Trial to Assess the Safety and Efficacy of Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-102-DED-031
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reproxalap Ophthalmic Solution (0.25%) (Experimental)
  Interventions: Drug: Reproxalap ophthalmic solution (0.25%)
- Vehicle Ophthalmic Solution (Placebo Comparator)
  Interventions: Drug: Vehicle ophthalmic solution

INTERVENTIONS:
Drug: Reproxalap ophthalmic solution (0.25%) — Reproxalap ophthalmic solution (0.25%) administered QID for four weeks, followed by BID administration for two weeks
  Arms: Reproxalap Ophthalmic Solution (0.25%)
Drug: Vehicle ophthalmic solution — Vehicle ophthalmic solution administered QID for four weeks, followed by BID administration for two weeks
  Arms: Vehicle Ophthalmic Solution

SUMMARY:
A Multicenter, Phase 3, Randomized, Double-Masked, Parallel-Group, Vehicle-Controlled, Environment Exposure Clinical Trial to Assess the Efficacy and Safety of 0.25% Reproxalap

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age;
* written informed consent and sign the Health Information Portability and Accountability Act (HIPAA) form;
* history of use or desire to use eye drops for dry eye symptoms within 6 months of Visit 1

Exclusion Criteria:

* ongoing ocular infection (bacterial, viral, or fungal) or active ocular inflammation at Visit 1;
* contact lenses within 7 days of Visit 1 or anticipate using contact lenses during the trial;
* eye drops within 2 hours of Visit 1;
* laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months;
* topical ocular cyclosporine, lifitegrast, corticosteroid, or any other topical ocular prescription medication within 90 days of Visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-11-03 (Actual); Study Completion 2024-11-03 (Actual)

PRIMARY OUTCOMES:
Subject-reported ocular discomfort score over Week 1 to Week 6 | From Day -14 to Day 43
  Measured using a 0 - 100 visual analog scale where 0 is "no discomfort" and 100 is "maximal discomfort"

CONTACTS AND LOCATIONS:
Locations (1):
- Core, Inc., Shelby, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No